CLINICAL TRIAL: NCT07117552
Title: Clinical and Radiological Pattern of Pleuropulmonary Affection in Patients With Connective Tissue Diseases
Brief Title: Study for Patients With Connective Tissue Diseases Who Suffer From Pleuropulmonary Symptoms Clinically and Radiologically
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrahman Amer Abdelwahab, Resident of chest department in sohag university hsopital, Sohag University
Other Study IDs: soh-med--25-7-3MS
Record Dates: First submitted 2025-08-01; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Connective Tissue Diseases
Keywords: Connective tissue diseases; Pulmonary affection; Pulmonary complications
MeSH Terms: conditions — Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study for clinical and radiological presentation of patients with connective tissue diseases who complain from pleuropulmonary symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients who have diagnosed as connective tissue disease Presented by pleuropulmonary affection

Exclusion Criteria:

* Patients who presented by pleuropulmonary affection due to disease other than connective tissue diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with connective tissue disease Presented by pleuropulmonary symptoms
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
assess clinical presentation and radiological pattern of pleuropulmonary affection in patients with connective tissue diseases, and evaluate their effect in outcome of connective tissue diseases | Day 1 admission

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt